CLINICAL TRIAL: NCT05351697
Title: An Open-label, Dose Escalation and Dose Expansion, Phase I Study of BR105 Injection to Evaluate the Safety, Tolerability and Antitumor Activity in Patients With Advanced Malignant Tumors
Brief Title: Clinical Study of BR105 Injection
Acronym: BR105-I
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company R&D Strategy Adjustment
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: BR105-I; CTR20220467 (Other: China Drug Trail); ChiCTR2200057711 (Other: China Clinical Tail Registry)
Record Dates: First submitted 2022-04-24; First posted 2022-04-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BR105 (Experimental): BR105 infusions will be administered weekly 21 days after the initial dose
  Interventions: Drug: BR105 injection

INTERVENTIONS:
Drug: BR105 injection — 0.2mg/kg, 1mg/kg, 3mg/kg, 10mg/kg, 20mg/kg, 30mg/kg, 40mg/kg respectively

SUMMARY:
A phase 1, dose escalation and dose expansion study of BR105 in patients with advanced malignancies.

DETAILED DESCRIPTION:
This phase 1 clinical study is an open-label, multiple-dose, dose-escalation, dose-expansion, safety, PK, PD study of BR105. The phase 1 protocol will have 2 parts: a single agent dose escalation phase (Part 1) and dose expansion phase (Part 2). Approximately 40-162 adult patients are expected to be enrolled in the study.

The starting dose for phase I is 0.2 mg/kg, followed by 6 dose cohorts (1, 3, 10, 20, 30 and 40 mg/kg). Duration of dose limiting toxicity (DLT) observation is 21 days. Each subject will receive an intravenous infusion of BR105 on day 1 and be observed for 21 days after a single dose. Then Each subject will receive BR105 weekly.

ELIGIBILITY:
Inclusion Criteria:

* 1. Be willing to sign the Informed Consent Form (ICF), and can follow the visit schedule and procedures defined in the protocol.
* 2. Male or female subject above 18 years old, no more than 75 years old.
* 3. Phase Ia only: Histologically/cytologically confirmed, subjects with advanced malignancies or recurrent or refractory malignant lymphoma， standard treatment failure or intolerance or no standard and effective treatment region. Phase Ib only: Subjects will be limited to specific subjects according to the results of phase Ia, and it is preliminarily proposed to be subjects with relapsed and refractory B-cell non-Hodgkin's lymphoma and advanced gastric cancer.
* 4. ECOG Performance Status 0 to 1.
* 5. Subjects with life expectancy of ≥ 3 months.
* 6. Phase Ia only: Subjects are not required to have measurable lesions at baseline, per RECIST v1.1 or Lugano 2014 criteria. Phase Ib only: Subjects must have at least one measurable lesion at baseline in phase Ib (bone metastasis or central nervous system (CNS) metastasis only is not accepted as a measurable lesion) , per RECIST v1.1 or Lugano 2014 criteria.
* 7. Any remaining toxicities from prior anti-tumor treatment should be restored to ≤ grade 1 as per CTCAE v5.0 or baseline level with exception of the residual hair loss.
* 8. Must have adequate organ and bone marrow function (except for subjects who use any cell factors, growth factors and blood transfusion treatment within 14 days before enrollment), inculding the following

  1. Neu≥ 1,500/mm3 (1.5×109/L)
  2. PLT ≥100,000/mm3（100×109/L）
  3. HGB ≥9g/dL（90g/L）
  4. Cr ≤1.5×ULN or Ccr ≥ 50 ml/min
  5. TBIL ≤1.5×ULN，subjects with liver metastasis or liver cancer ≤2×ULN
  6. AST or ALT ≤2.5×ULN, subjects with liver metastasis or liver cancer≤5×ULN
  7. INR ≤1.5， PT and APTT ≤1.5×ULN
* 9. Female subjects of child-bearing potential must enter the study with a negative serum pregnancy test result. Female subjects of child-bearing potential or male subjects with female partners of child-bearing potential must be willing to use viable contraception method that is deemed effective by the investigator throughout the treatment period and for at least 6 months following the last dose of study drug

Exclusion Criteria:

* 1. Subjects with known allergy to the test drug or any of its excipients, or severe allergic reaction to other monoclonal antibodies.
* 2. Prior treatment with CD47 or signal regulatory protein alpha-targeting agents.
* 3. History of hemolytic anemia (including Evans syndrome) or autoimmune thrombocytopenia caused by any reason within 3 months before the first administration of the test drug.
* 4. Subjects who are receiving thrombolytic or anticoagulant therapy due to high risk of thrombosis.
* 5. Received the following treatments or drugs before the first study treatment.

  1. Subjects who have had major surgery within the 28-days from the first dosing, or plan to have major surgery during the study (tissue biopsy due to diagnosis is allowed).
  2. Subjects who have received immunosuppressive drugs within the 28-days from the first dosing; Subjects can receive nasal and inhaled corticosteroids or physiological doses of systemic steroid hormones (i.e. ≤ 10mg/day prednisone or other corticosteroids with equivalent pharmacological doses) in the absence of active autoimmune diseases.
  3. Subjects who have received live attenuated vaccine within 28 days before the first dosing, or who plan to receive during the study and within 60 days after the last dosing.
  4. Subjects who have received anti-tumor treatments (including chemotherapy, radiotherapy, immunotherapy, endocrine therapy, targeted therapy, biotherapy or tumor embolization) within 28 days before the first dosing, or used therapeutic radiopharmaceuticals within 56 days before the first trial drug treatment.
  5. Subjects who have participated in other clinical trials and used trial related drugs within 28 days before the first dosing.
* 6. Subjects with a history of active autoimmune diseases or autoimmune diseases that may recur, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel diseases, Hashimoto's thyroiditis, etc., with exception of alternative treatment requirements (such as residual hypothyroidism caused by autoimmune thyroiditis).
* 7. Subjects with metastatic cancer of central nervous system, uncontrollable pleural effusion, pericardial effusion or peritoneal effusion (except for subjects with indwelling catheter); Or subjects with uncontrollable hypercalcemia; Or subjects with spinal cord compression.
* 8. Subjects with any other malignancies in the past 2 years, excluding fully cured cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin, other malignancies that have been treated in the past and the current disease condition is stable, and other malignancies may benefit from this trial based on judgements of investigators.
* 9. Positive for human immunodeficiency virus (HIV) antibody. Positive for treponema pallidum (TP) antibody. Positive for hepatitis C virus (HCV) antibody, and HCV RNA≥ the lower limit of detection. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb), and HBV DNA ≥ 1ⅹ103IU/ml.
* 10. Subjects with severe poorly controlled concomitant diseases, such as congestive heart failure (NYHA grade II or above), arrhythmias or angina pectoris that increase thromboembolic events, coronary artery stenting, angioplasty or coronary artery bypass grafting in recent 6 months, uncontrolled hypertension after treatment (systolic blood pressure ≥ 160mmhg or diastolic blood pressure ≥ 100mmhg), etc.
* 11. Subjects with history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; If immunosuppressive transplantation is not required, it can be included (such as corneal transplantation and hair transplantation).
* 12. Subjects with any active infection requiring systemic treatment by intravenous infusion occurred within 14 days before enrollment.
* 13. Subjects who have active tuberculosis, or have received anti-tuberculosis treatment within 1 year prior to screening.
* 14. Subjects with interstitial lung diseases, such as interstitial pneumonia, pulmonary fibrosis, or non-infectious pneumonia.
* 15. Subjects who have suffered from diseases affecting intravenous infusion and venous blood collection currently.
* 16. Subjects with known or suspected non-compliance with study protocol (e.g. psychotropic substance abuse, alcohol dependence, psychological disorder or drug abuse history).
* 17. Pregnant or breastfeeding women.
* 18. Subjects who, in the judgment of the investigator, are not suitable for enrollment or may not be able to complete the experiment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) (Phase Ia) | Up to 3 weeks
  Number of subjects with a DLT
Maximum tolerated dose (MTD) (Phase Ia) | Up to 3 weeks
  Determine maximum tolerated dose (MTD) of BR105
Number of subjects with adverse events (Phase Ia) | Up to 12 mouths
  Number of subjects who experienced an adverse event
Objective response rate (ORR) (Phase Ib) | Up to 2-3 years
  Phase Ib, BR105 Antitumor Activity (ORR)
Recommended phase 2 dose (RP2D) (Phase Ib) | Up to 2-3 years.
  Determine recommended phase 2 dose (RP2D) of BR105.

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of BR105 (Phase Ia and Phase Ib ) | Up to 12 mouths for Phase Ia; Up to 2-3 years for Phase Ib
  To determine the maximum serum concentration (Cmax) of BR105
Time of Maximum observed serum concentration (Tmax) of BR105 (Phase Ia and Phase Ib ) | Up to 12 mouths for Phase Ia; Up to 2-3 years for Phase Ib
  To determine the Tmax of BR105.
Serum Half-life (T-HALF) of BR105.(Phase Ia and Phase Ib ) | Up to 12 mouths for Phase Ia; Up to 2-3 years for Phase Ib
  To determine the t1/2 of BR105.
Objective response rate (ORR) (Phase Ia ) | Up to 12 mouths for Phase Ia
  Number of participants who achieved a best response of either complete response (CR) or partial response (PR) during treatment evaluated by investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Lugano 2014.
Progression free survival (PFS)(Phase Ia and Phase Ib ) | Up to 12 mouths for Phase Ia; Up to 2-3 years for Phase Ib
  To determine the PFS by investigator.
Number of patients with adverse events (Phase Ia and Phase Ib ) | Up to 12 mouths for Phase Ia; Up to 2-3 years for Phase Ib
  Incidence of AE as assessed by CTCAE 5.0
Immunogenicity (Phase Ia and Phase Ib ) | Up to 12 mouths for Phase Ia; Up to 2-3 years for Phase Ib
  Anti-Drug Antibodies (ADA) will be tested and percentage of ADA positive patients will be calculated to evaluate immunogenicity of BR105

OTHER OUTCOMES:
Biomarker | Up to 12 mouths
  SIRPα levels and percentage of SIRPα receptor occupancy in peripheral blood CD14+ monocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China